CLINICAL TRIAL: NCT03505255
Title: Comparison Between Intraperitoneal Versus Intramuscular Neostigmine on Pattern of Postoperative GIT Motility in Patients Undergoing Laparoscopic Cholecystectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Haitham Mohammad Ahmad Mohammad, Doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GIT motility after lap.
Record Dates: First submitted 2018-04-05; First posted 2018-04-23 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Pattern of GIT Motility
MeSH Terms: interventions — Neostigmine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Active Comparator): Group A: 40 patients will receive intraperitoneal neostigmine 0.25 mg in 30 ml normal saline and 1 ml normal saline intramuscular.
  Interventions: Drug: Neostigmine
- Group B (Active Comparator): Group B: 40 patients will receive intraperitoneal neostigmine 0.5 mg in 30 ml normal saline and 1 ml normal saline intramuscular.
  Interventions: Drug: Neostigmine
- Group C (Active Comparator): Group C: 40 patients will receive intramuscular neostigmine 0.5 mg in 1 ml volume plus 30 ml normal saline intraperitoneal.
  Interventions: Drug: Neostigmine
- Group D (Placebo Comparator): Group D (control group): 40 patients will receive intraperitoneal 30 ml normal saline and 1 ml normal saline intramuscular.
  Interventions: Other: Normal saline

INTERVENTIONS:
Drug: Neostigmine — Neostigmine is a cholinesterase-inhibitor, which augments the concentration of acetylcholine (ACh) at the neuromuscular junction
  Arms: Group A; Group B; Group C
Other: Normal saline — Normal saline 0.9 % is given in the control group
  Arms: Group D

SUMMARY:
The goal in this work is to compare between the effects of intraperitoneal versus intramuscular neostigmine on pattern of postoperative GIT motility in patients undergoing laparoscopic cholecystectomy

DETAILED DESCRIPTION:
Despite numerous advances in surgical technique and perioperative care, postoperative ileus (POI) continues to be one of the most common and expected aspects of abdominal surgery. It prolongs hospital stays, increases medical costs and frustrates patients and surgeons.

Many authors suggest that POI is a mandatory phase of the recovery period for any intra-abdominal procedure, and only an ileus lasting greater than 5 days is abnormal - to be termed a prolonged POI.

Under this definition, fully 40% of patients undergoing laparotomy experience prolonged postoperative ileus.

In 2006, different types of postoperative ileus (primary, secondary, recurrent, prolonged) were defined through consensus, and prolonged postoperative ileus was defined as absence of bowel function after the third postoperative day for laparoscopic surgery and after the fifth postoperative day for open abdominal surgery.

What constitutes prolonged postoperative ileus is debated, with many different definitions reported; consequently reported incidences range from 3% to 32%. Neostigmine is a cholinesterase-inhibitor, which augments the concentration of acetylcholine (ACh) at the neuromuscular junction, thereby increasing contractions in the normal gut.

ELIGIBILITY:
Inclusion Criteria:

ASA status I and II patients, aged between 20 and 60 years, who are scheduled for laparoscopic cholecystectomy.

-

Exclusion Criteria:

Patients with electrolyte imbalance Patients with diabetes mellitus Patients who are addict to opioids Patients with neurological defects or paralysis or preoperative recumbence. Patients with atrial-ventricular conduction disturbances, sinus bradycardia < 60 BPM or a nodal rhythm.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
passing flatus | each 2 hours
  A questionnaire for each patient about the first time to pass flatus or stool

SECONDARY OUTCOMES:
Barium meal | after 4 hours, 24hours, 48 hours
  Upon regaining consciousness in the recovery room after operation, the patient will be asked to swallow another 30 cc. of liquid barium and 4 hours later abdominal roentgenogram film will be taken.

REFERENCES:
- [Background] Baig MK, Wexner SD. Postoperative ileus: a review. Dis Colon Rectum. 2004 Apr;47(4):516-26. doi: 10.1007/s10350-003-0067-9. Epub 2004 Feb 25. PMID 14978625 (Retraction: PMID 16132474 Wexner SD. Dis Colon Rectum. 2005 Oct;48(10):1983; PMID 16132475 Dis Colon Rectum. 2005 Oct;48(10):1983)
- [Background] Delaney CP, Wolff BG, Viscusi ER, Senagore AJ, Fort JG, Du W, Techner L, Wallin B. Alvimopan, for postoperative ileus following bowel resection: a pooled analysis of phase III studies. Ann Surg. 2007 Mar;245(3):355-63. doi: 10.1097/01.sla.0000232538.72458.93. PMID 17435541
- [Background] Schuster R, Grewal N, Greaney GC, Waxman K. Gum chewing reduces ileus after elective open sigmoid colectomy. Arch Surg. 2006 Feb;141(2):174-6. doi: 10.1001/archsurg.141.2.174. PMID 16490895
- [Background] Sajja SB, Schein M. Early postoperative small bowel obstruction. Br J Surg. 2004 Jun;91(6):683-91. doi: 10.1002/bjs.4589. PMID 15164435
- [Background] Viscusi ER, Goldstein S, Witkowski T, Andonakakis A, Jan R, Gabriel K, Du W, Techner L, Wallin B. Alvimopan, a peripherally acting mu-opioid receptor antagonist, compared with placebo in postoperative ileus after major abdominal surgery: results of a randomized, double-blind, controlled study. Surg Endosc. 2006 Jan;20(1):64-70. doi: 10.1007/s00464-005-0104-y. Epub 2005 Dec 7. PMID 16333556
- [Background] Husebye E. Gastrointestinal motility disorders and bacterial overgrowth. J Intern Med. 1995 Apr;237(4):419-27. doi: 10.1111/j.1365-2796.1995.tb01196.x. PMID 7714466
- [Background] Holte K, Kehlet H. Postoperative ileus: a preventable event. Br J Surg. 2000 Nov;87(11):1480-93. doi: 10.1046/j.1365-2168.2000.01595.x. PMID 11091234
- [Background] Goyal RK, Hirano I. The enteric nervous system. N Engl J Med. 1996 Apr 25;334(17):1106-15. doi: 10.1056/NEJM199604253341707. No abstract available. PMID 8598871